CLINICAL TRIAL: NCT00950495
Title: Effects of an Oral Appliance on Obstructive Sleep Apnea: A Randomized, Placebo-Controlled Trial
Brief Title: Oral Appliance Therapy in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Ghizlane Aarab, Dr., VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U/1731/0326
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Parallel design; Oral appliance; Mandibular advancement device; Continuous positive airway pressure; Placebo; Therapy; Side-effects; Compliance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mandibular advancement device (MAD) (Active Comparator): an MAD is placed in the mouth prior to sleep. After waking up in the morning, the appliance is removed.
  Interventions: Device: Mandibular Advancement Device (MAD)
- nasal CPAP (Active Comparator): The device is turned on, and the nasal mask is placed on the nose prior to sleep. After waking up in the morning, the device is turned off and the mask is removed
  Interventions: Device: nasal CPAP
- placebo (Placebo Comparator): the placebo appliance is placed in the mouth prior to sleep. After waking up in the morning, the appliance is removed.
  Interventions: Device: placebo

INTERVENTIONS:
Device: Mandibular Advancement Device (MAD) — This oral appliance keeps the mandible and the tongue in a protruded position. This results in an upper respiratory tract widening and/or reduced collapsibility of the upper airway, thereby preventing the upper airway collapse during sleep.
  Other Names: mandibular repositioning appliance; mandibular advancement appliance; mandibular repositioning device; mandibular repositioning splint; mandibular advancement splint; oral appliance
  Arms: Mandibular advancement device (MAD)
Device: nasal CPAP — The CPAP machine delivers a stream of compressed air via a hose to a nose mask, splinting the airway (keeping it open under air pressure) so that unobstructed breathing becomes possible, reducing and/or preventing apneas and hypopneas
  Arms: nasal CPAP
Device: placebo — as a placebo, a thin (< 1 mm), hard acrylic-resin palatal splint with only a partial palatal coverage was used
  Arms: placebo

SUMMARY:
The aim of the study was to compare the effects of a mandibular advancement device (MAD) with those of nasal continuous positive airway pressure(nCPAP) and of an intra-oral placebo device in obstructive sleep apnea (OSA) patients. The hypothesis for this study was that both MAD therapy and nCPAP therapy have similar, better treatment effects than placebo therapy in OSA. The study was performed according to the CONSORT (consolidated standards of reporting trials) statement (Altman et al., 2001), employing a parallel-group, randomized, placebo-controlled trial design.

DETAILED DESCRIPTION:
Setting and participants:

Eligible OSA patients, living in the greater Amsterdam area, were referred to the Slotervaart Medical Center by their family physician. All patients underwent a thorough medical examination, including a full polysomnographic (PSG) recording, at the departments of Neurology, Pulmonary Medicine, and ENT, as well as a thorough dental examination at the Department of Oral Kinesiology of ACTA. OSA patients were invited for participation in this study when they fulfilled the inclusion criteria and exclusion criteria.

Randomisation and allocation:

After written informed consent was obtained, the patients were randomly allocated to one of three therapy groups (MAD, nCPAP, or placebo; see below). To ensure that the groups were of approx. the same size, block randomisation was used. Block sizes were 6, 12, and 18; sizes were randomly varied. The allocation sequence was automatically generated and subsequently concealed by an independent co-worker, who kept a paper copy in a lockable drawer. Sealed opaque envelopes were used to conceal the allocation from the principal investigator.

Interventions and blinding:

Three forms of therapy interventions were used in this parallel-group study. First, an individually fabricated MAD with an adjustable protrusive mandibular position at a constant vertical dimension was used. Second, nCPAP of the REMstar Pro system was used (Respironics, Herrsching, Germany). Third, a thin (< 1 mm), hard acrylic-resin palatal splint with only a partial palatal coverage was used as a placebo.

Patients were blinded to the nature of the assigned therapy (placebo or active). After evaluating the therapy, all patients were asked if they were of the opinion that they had received an active or placebo treatment. Blinding of the analyst was ascertained by assigning codes to data sets and by analyzing these sets in random blocks.

Procedure:

From all patients, two full polysomnographic (PSG) recordings were obtained in the sleep laboratory of the Slotervaart Medical Center, using Siesta hardware and Pro-Fusion software (Compumedics, Abbotsford, Australia): one before therapy assignment (baseline PSG) and one after 6 ± 2 months (mean ± SD) of treatment (therapy evaluation PSG). For the MAD and nCPAP groups, the third and fourth PSG recordings for therapy evaluation were performed 6 months and one year after the first therapy evaluation (long-term follow-up). The primary and secondary outcome measures were obtained at baseline and at therapy evaluations.

The MAD and nCPAP were titrated before the start of the treatment. The titration of the nCPAP was performed during a third sleep laboratory examination. The pressure was increased in incremental steps of 1 cm H2O/h, until respiratory disturbances and respiration-related arousals were reduced to ≤ 5/h, and snoring was minimized.

For the titration of the MAD, four ambulatory PSG recordings were obtained at regular intervals, using Monet hardware and Rembrandt Software (Medcare Automation B.V., Amsterdam, The Netherlands). The most effective protrusion position of the MAD (i.e., the mandibular position that yielded the lowest AHI value) was chosen from among four randomly offered positions (viz., 0%, 25%, 50%, and 75% of the maximum protrusion).

For the placebo group, the study procedure was made equally intense as that for the MAD group by making four ambulatory PSG recordings at regular intervals as well.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* apnea-hypopnea index (AHI) between 5 and 45 events per hour

Exclusion Criteria:

* evidence of respiratory/ sleep disorders other than obstructive sleep apnea
* a body mass index (BMI) > 40
* medication usage that could influence respiration or sleep
* periodic limb movement disorder
* previous treatment with CPAP or MAD
* reversible morphological upper airway abnormalities (e.g., enlarged tonsils)
* temporomandibular disorders (based on a functional examination of the masticatory system)
* untreated periodontal problems
* dental pain
* lack of retention possibilities for a mandibular advancement device or a placebo appliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-10; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index (AHI) | 6 months

SECONDARY OUTCOMES:
other respiratory variables (apnea-hypopnea index during different sleep stages and positions);sleep variables (sleep stages and arousals);excessive daytime sleepiness;health perception;compliance;snoring reports; side-effects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ghizlane Aarab, DDS, Principal Investigator — Academic Centre for Dentistry Amsterdam (ACTA), Research Institute Move, University of Amsterdam and VU University Amsterdam
Locations (1):
- Academic Centre for Dentistry Amsterdam (ACTA), Research Institute Move, University of Amsterdam and VU University Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Result] Aarab G, Lobbezoo F, Hamburger HL, Naeije M. Effects of an oral appliance with different mandibular protrusion positions at a constant vertical dimension on obstructive sleep apnea. Clin Oral Investig. 2010 Jun;14(3):339-45. doi: 10.1007/s00784-009-0298-9. Epub 2009 Jun 18. PMID 19536571
- [Result] Aarab G, Lobbezoo F, Hamburger HL, Naeije M. Variability in the apnea-hypopnea index and its consequences for diagnosis and therapy evaluation. Respiration. 2009;77(1):32-7. doi: 10.1159/000167790. Epub 2008 Oct 29. PMID 18957843
- [Result] Aarab G, Lobbezoo F, Wicks DJ, Hamburger HL, Naeije M. Short-term effects of a mandibular advancement device on obstructive sleep apnoea: an open-label pilot trial. J Oral Rehabil. 2005 Aug;32(8):564-70. doi: 10.1111/j.1365-2842.2005.01467.x. PMID 16011634
- [Result] Aarab G, Lobbezoo F, Hamburger HL, Naeije M. Oral appliance therapy versus nasal continuous positive airway pressure in obstructive sleep apnea: a randomized, placebo-controlled trial. Respiration. 2011;81(5):411-9. doi: 10.1159/000319595. Epub 2010 Oct 20. PMID 20962502
- [Result] Aarab G, Lobbezoo F, Heymans MW, Hamburger HL, Naeije M. Long-term follow-up of a randomized controlled trial of oral appliance therapy in obstructive sleep apnea. Respiration. 2011;82(2):162-8. doi: 10.1159/000324580. Epub 2011 Mar 31. PMID 21454959
- [Result] Nikolopoulou M, Naeije M, Aarab G, Hamburger HL, Visscher CM, Lobbezoo F. The effect of raising the bite without mandibular protrusion on obstructive sleep apnoea. J Oral Rehabil. 2011 Sep;38(9):643-7. doi: 10.1111/j.1365-2842.2011.02221.x. Epub 2011 Apr 5. PMID 21463349